CLINICAL TRIAL: NCT03189355
Title: Expression of Protein Tyrosine Phosphatase 1B (PTP1B) and Body Composition Modification in Patients With Septic Shock
Acronym: Coc-SEPP1B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016/108/HP
Record Dates: First submitted 2017-05-22; First posted 2017-06-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients With Septic Shock (Experimental): Blood sampling on D1 PTP1B + zonulin +PAXGENE tube +aprotinin tube and D4 zonulin Bioelectrical impedance vector analysis on D1 + D4 Muscular echography on D1 + D4
  Interventions: Procedure: Blood sampling; Procedure: Bioelectrical impedance vector analysis; Procedure: Muscular echography

INTERVENTIONS:
Procedure: Blood sampling — * D1 PTP1B + zonulin +PAXGENE tube +aprotinin tube
  * D4 zonulin
Procedure: Bioelectrical impedance vector analysis — * D1
  * D4
Procedure: Muscular echography — * D1
  * D4

SUMMARY:
With a prevalence of more than 15% in ICU, septic shock today represents a real public health problem and remains the leading cause of mortality in ICU. Undernutrition is characterized by an alteration of the body composition and in particular by a loss of muscle mass. In intensive care, there are indirect elements suggesting a link between loss of muscle mass and prognosis.

Muscle mass results from a balance between the pathway of proteolysis and that of protein synthesis, depending on many factors, not one of the most important are insulin. The protein PTP1B (Protein Tyrosine Phosphatase 1B), by the dephosphorylation of its numerous substrates, constitutes an endogenous regulator of numerous intracellular signaling pathways, including that of insulin. PTP1B could play a role in the protein synthesis abnormalities observed during sepsis leading clinically to impaired body composition including muscle body mass. Therefore, we propose to study the association between PTP1B and loss of muscle mass in patients in sepsis in resuscitation.

The intestinal barrier plays an essential role in protecting against microbial luminal flora and the phenomenon of bacterial translocation. Zonulin is one of the major regulators of tight junctions, important actors in the intestinal barrier function. The increase in plasma zonulin levels, greater than 0.6 ng / mg, is directly correlated with increased intestinal permeability (16). However, elevation of plasma zonulin has never been evaluated in septic resuscitation patients. This is why we propose the evaluation of the association between plasma zonulin and the loss of muscle mass in these resuscitation patients.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock or severe sepsis
* Age > 18 years old
* Affiliation to a social security system
* Information and consent. If patient cannot give his consent, an emergency consent will be sign by trusted person
* Contraception for woman, of childbearing age

Exclusion Criteria:

* Pregnancy or breastfeeding
* Prisoners
* Patient with pacemaker or defibrillator
* patient participating to a clinical trial with the same primary outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
PTP1B analysis | Day 1
  1 PAXgene tube (2,5 ml) will be used. RNA extraction will be done with a PAXgene Blood RNA System kit.
Muscular composition | Day 1
  Muscular composition will be measured by muscular echography with a 2B mode on D1 and D4 from the admission.T
Muscular composition | Day 4
  Muscular composition will be measured by muscular echography with a 2B mode on D1 and D4 from the admission.T

SECONDARY OUTCOMES:
Intestinal permeability | Day 1
  1 tube of 5 ml Aprotinin will be taken on D1 and D4 to determine the expression of plasma zonulin. The concentration will be assayed by ELISA using a commercial kit (MyBiosource, USA).
Intestinal permeability | Day 4
  1 tube of 5 ml Aprotinin will be taken on D1 and D4 to determine the expression of plasma zonulin. The concentration will be assayed by ELISA using a commercial kit (MyBiosource, USA).
Body composition | Day 1
  Body composition will be measured by impedancemetry on D1 and D4
Body composition | Day 4
  Body composition will be measured by impedancemetry on D1 and D4

CONTACTS AND LOCATIONS:
Overall Officials: Caroline LEMAITRE, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No